CLINICAL TRIAL: NCT03706261
Title: Alzheimer's PET Imaging in Racially/Ethnically Diverse Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adam Brickman (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Adam Brickman, Associate Professor of Neuropsychology, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AAAR8986; 1RF1AG058067-01A1 (NIH)
Record Dates: First submitted 2018-10-11; First posted 2018-10-15 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease
Keywords: Tau; Amyloid; MK-6240; Florbetaben; Racial/Ethnic Minority; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease; Pick Disease of the Brain | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Offspring Cohort (Experimental): Racially/ethnically diverse subjects with or without a positive family history of Alzheimer's disease (AD) will have one PET scan with 18F-MK-6240 over a 30 to 60-minute scanning period, and one PET scan with 18F-Florbetaben over a 20-minute scanning period.
  Interventions: Drug: 18F-MK-6240; Drug: 18F-Florbetaben

INTERVENTIONS:
Drug: 18F-MK-6240 — Administration of 5 mCi of 18F-MK-6240 for tau PET.
  Other Names: [18F]MK-6240
Drug: 18F-Florbetaben — Administration of 8.1 mCi as a slow single intravenous bolus (6 sec/mL) in a total volume of up to 10 mL of 18F-Florbetaben for Aβ PET imaging.
  Other Names: [18F]Florbetaben

SUMMARY:
The study employs tau positron emission tomography (PET) imaging in a well-characterized multi-racial/ethnic cohort to examine the extent to which tau pathology is associated with cognition, differences in tau pathology across racial/ethnic groups, and the relationship between MRI markers of small-vessel cerebrovascular disease and tau pathology. The study also investigates amyloid-dependent tau spreading.

DETAILED DESCRIPTION:
Deposition of hyperphosphorylated tau protein is observed in several neurodegenerative diseases including Alzheimer's Disease (AD), progressive supranuclear palsy, corticobasal degeneration, chronic traumatic encephalopathy, and frontotemporal lobar degeneration. Tau is a microtubular protein and its native function is to provide structural support to neurons. Paired helical filaments composed of dysfunctional tau protein are found in several neurodegenerative diseases. In AD, the clinical progression of dementia has been shown to correlate with the amount and topographical spread of tau throughout the brain. Therefore, detecting and quantifying tau aggregate load in brain would have diagnostic and prognostic potential in clinical management of several neurological diseases. As disease modifying drugs that target tau are being developed, there is a critical need for a reliable method of detecting tau aggregates to confirm pathology in patients entering clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35 - 85 years
* Have either mild cognitive impairment or mild clinical Alzheimer's disease; or have no problem with memory or thinking.
* Able to participate in all scheduled evaluations and to complete all required tests and procedures
* Considered likely to comply with the study protocol and to have a high probability of completing the study

Exclusion Criteria:

* Past or present history of a certain brain disease other than mild cognitive impairment or mild clinical Alzheimer's disease.
* Certain significant medical conditions. Examples are uncontrolled epilepsy or multiple serious injuries.
* Unable to lie still for PET scans.
* Radiation exposure for research studies in the last year that would put you past allowable limits if included in this study.
* Participation in the last year in a clinical trial for a disease modifying drug for AD unless it can be determined that your received placebo and not active drug.
* Conditions that preclude entry into the scanner (e.g. claustrophobia, etc.).
* Inability to have a catheter in your vein for the injection of the radioligand (dye).
* Currently pregnant or breastfeeding.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam M. Brickman, Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Analyses are planned to be on the group level. However, we may emphasize cases that are interesting on the individual level.

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Racially/ethnically diverse subjects with or without a positive family history of Alzheimer's disease (AD) will have one PET scan with 18F-MK-6240 over a 30 to 60-minute scanning period, and one PET scan with 18F-Florbetaben over a 20-minute scanning period.
Period: Overall Study
Arm/Group | All Participants
Started | 145
Completed | 126
Not Completed | 19

BASELINE CHARACTERISTICS:
Population: Of the 145 participants who consented to be in the study, 3 participants withdrew prior to receiving any scan. No baseline data was collected from these 3 participants.
Arm/Group | All Participants
Number analyzed (Participants) | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 106
  >=65 years | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 71
  Not Hispanic or Latino | 71
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 48
  White | 23
  More than one race | 0
  Unknown or Not Reported | 71
Region of Enrollment [Number; unit: participants]
  United States | 142

OUTCOME MEASURES:

1. Primary Outcome: Regional SUVR Value for 18F-MK-6240
Description: Regional standardized uptake value ratio (SUVR) for 18F-MK-6240 will be calculated to investigate associations with measures of memory, olfactory function, and cerebrovascular disease.
Time Frame: 1 day
Population: 115 participants had complete PET scans with this tracer
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | All Participants
Number analyzed (Participants) | 115
SUVR | 1.27 (0.23)

2. Primary Outcome: Number of Participants With Amyloid Positivity (Aβ+) for 18F-Florbetaben
Description: 18F-Florbetaben will be calculated to investigate the potential moderation of amyloid on the associations with tau.
Time Frame: 1 day
Population: 126 participants had complete PET scans with this tracer
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 126
Participants | 12

ADVERSE EVENTS:
Time Frame: 1 day for each scan, within 24 months of each other
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/142
Serious Adverse Events (participants affected / at risk) | 0/142
Other Adverse Events (participants affected / at risk) | 19/142
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=142)
Headache (General disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT03706261/Prot_SAP_000.pdf